CLINICAL TRIAL: NCT06865170
Title: Pain Perception During Intra-Articular Knee Joint Injection: What is the Effect of Needle Gauge and the Use of Ethyl Chloride?
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2200055
Record Dates: First submitted 2025-02-13; First posted 2025-03-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis (OA) of the Knee; Fear of Needles
Keywords: pain perception; fear of needles; needle gauge; ethyl chloride; corticosteroid injection; 25G versus 22G
MeSH Terms: conditions — Osteoarthritis; Iatrophobia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 22 Gauge Needle WITH Ethyl Chloride spray (Experimental): This group will receive an intra-articular knee joint injection using a 22 gauge needle, and will be pre-anesthetized with ethyl chloride spray
  Interventions: Procedure: 22 gauge needle; Procedure: +/- Ethyl Chloride Topical Aerosol Anesthetic
- 25 Gauge Needle WITH Ethyl Chloride spray (Experimental): This group will receive an intra-articular knee joint injection using a 25 gauge needle, and will be pre-anesthetized with ethyl chloride spray
  Interventions: Procedure: 25 gauge needle; Procedure: +/- Ethyl Chloride Topical Aerosol Anesthetic
- 22 Gauge Needle WITHOUT Ethyl Chloride spray (Placebo Comparator): This group will receive an intra-articular knee joint injection using a 22 gauge needle, and will be pre-anesthetized with a PLACEBO spray
  Interventions: Procedure: 22 gauge needle; Procedure: +/- Ethyl Chloride Topical Aerosol Anesthetic
- 25 Gauge Needle WITHOUT Ethyl Chloride spray (Placebo Comparator): This group will receive an intra-articular knee joint injection using a 25 gauge needle, and will be pre-anesthetized with a PLACEBO spray
  Interventions: Procedure: 25 gauge needle; Procedure: +/- Ethyl Chloride Topical Aerosol Anesthetic

INTERVENTIONS:
Procedure: 25 gauge needle — This intervention will observe patients post-procedural pain using a 25 gauge needle
  Arms: 25 Gauge Needle WITH Ethyl Chloride spray; 25 Gauge Needle WITHOUT Ethyl Chloride spray
Procedure: 22 gauge needle — This intervention will observe patients post-procedural pain using a 22 gauge needle
  Arms: 22 Gauge Needle WITH Ethyl Chloride spray; 22 Gauge Needle WITHOUT Ethyl Chloride spray
Procedure: +/- Ethyl Chloride Topical Aerosol Anesthetic — This intervention will observe patients post-procedural pain when using topical ethyl chloride spray. This will be compared to a placebo spray which will utilize isopropyl alcohol.

SUMMARY:
This study aims to investigate factors that affect the subjective experience of pain during and after intra-articular knee joint injection of steroids by comparing needle gauge size (22 G vs 25 G needles), as well as the presence or absence of topical ethyl chloride spray. Additionally, this study will investigate the effects of other various factors on patients' pain associated with the injection. Lastly, this study aims to determine the effect of patients' subjective pain from the injection on long-term clinical outcomes.

Specific aims are as follows:

Aim 1): Determine the effect of needle gauge size on patient reported pain associated with an ultrasound-guided intra-articular knee injection.

Aim 2): Determine the effect of ethyl chloride spray on patient reported pain associated with an ultrasound-guided intra-articular knee injection.

Aim 3): Determine the effect of sex, age, BMI, thigh size, severity of OA, and fear of needles on patient pain associated with an ultrasound-guided intra-articular knee injection.

Aim 4) Determine the effect of patient pain from the procedure on longer term clinical outcomes after an ultrasound-guided intra-articular knee steroid injection.

Researchers will obtain data at various time points, including pre-procedural data, immediately after the procedure, 24-48 hours after, and 6 weeks post-procedure.

Participants will:

Consent to receiving an intra-articular knee joint injection with steroids if indicated.

Score their "procedural" pain immediately following the procedure, score their post-procedural "soreness" 24-48 hours after via telephone call, and score their overall knee pain about 6 weeks after the procedure via telephone call.

DETAILED DESCRIPTION:
Hypotheses to be tested:

Hypothesis 1): Patients who receive an ultrasound-guided intra-articular knee steroid injection with a 25G needle will report less pain from the procedure at the time of the procedure and less procedure-related pain 24-48 hours after the procedure

Hypothesis 2) Patients who receive an ultrasound-guided intra-articular knee steroid injection with use of ethyl chloride with a given needle gauge will report less pain from the procedure at the time of the procedure and 24-48 hours after the procedure

Hypothesis 3) Higher thigh circumference and fear of needles will be associated with higher levels of pain from the procedure at the time of the procedure and 24-48 hours after the procedure

Hypothesis 4) Higher levels of patient pain during the injection procedure will be associated with lower improvements in knee osteoarthritis pain and knee functional scores at 6 weeks.

There is evidence to suggest that by effectively altering certain parameters and techniques such as needle gauge diameter, speed of administration, and angle of needle during subcutaneous injection of local anesthetic, one can effectively improve the subjective experience of the patient. Evidence also suggests that choice of needle gauge size - which is at the discretion of the practitioner - may be inversely proportional to patient's perception of pain during an injection procedure. Topical anesthesia, such as via the use of ethyl chloride spray (which is also at the discretion of the practitioner), may also modify procedural pain. Furthermore, some studies suggest a correlation between patients' pain during a procedure and their clinical outcomes from the injection.

However, the current research is primarily composed of studies investigating subcutaneous injections (e.g. insulin or vaccination injections) using relatively small needle gauges, or of anesthetic injections in the spine. As such, there is very limited research on factors which may impact peripheral joint injections. Furthermore, there is a paucity of information regarding the effect of patient factors such as age, sex, limb size, anxiety, and fear of needles on the perception of pain during peripheral intra-articular injections.

Additional knowledge regarding the use of different needle gauge and/or the use of local anesthetic may help guide physician treatment patterns with the goal of optimizing patient satisfaction. Additionally, by obtaining subjective data at multiple time points, including 6 weeks post-injection, investigators hope to determine if differences in patient experience with the procedure is associated with patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 40 years
2. fulfillment of the American College of Rheumatology criteria for knee OA
3. confirmation of knee-related pain and/or functional loss by clinical examination.
4. Patients with either

   1. bilateral knee OA/injections, or
   2. unilateral knee OA/injections.
5. Agreed to an intra-articular knee joint injection with steroids
6. Naive to use of ethyl chloride

Exclusion Criteria:

1. Arthroscopy of the index knee(s) within the prior 6 months
2. Steroid injection of the knee(s) within the prior 3 months
3. Hyaluronic acid or platelet-rich plasma injection of the knee within the prior 6 months
4. Patient reported prior injection of any type with ethyl chloride spray
5. Knee effusion requiring aspiration at the time of the procedure
6. Cognitively impaired individuals

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
NRPS for injection-related pain at the time of the procedure | immediately following the procedure
  NRPS = "Numeric Rating of Pain Scale", scale from 0 to 100. "0" = minimum score, better outcome); "100" (maximum score, worse outcome)

SECONDARY OUTCOMES:
NRPS pain 24-48 hours after the procedure at the injection site, assessing injection-related "soreness" | 28-48 hours after the procedure
  NRPS = "Numeric Rating of Pain Scale", scale from 0 to 100. "0" = minimum score, better outcome); "100" (maximum score, worse outcome)
NPRS score for overall knee pain, and WOMAC functional scores at six weeks post-procedure | 6 weeks following procedure
  NRPS = "Numeric Rating of Pain Scale", scale from 0 to 100. "0" = minimum score, better outcome); "100" (maximum score, worse outcome).
  WOMAC = "Western Ontario and McMaster Universities Arthritis Index" is a self-administered questionnaire consisting of 24 items divided into 3 subscales. Test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Sports Medicine Clinic, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided